CLINICAL TRIAL: NCT02049541
Title: A Phase I Study of BKM120 and Rituximab in Patients With Relapsed or Refractory Indolent B-Cell Lymphoma
Brief Title: Study of BKM120 & Rituximab in Patients With Relapsed or Refractory Indolent B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kami Maddocks, MD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Kami Maddocks, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13027; NCI-2014-00110 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
Keywords: BKM120; B-Cell Lymphoma; PI3K inhibitor
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell | interventions — NVP-BKM120; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PI3K inhibitor BKM120, rituximab) (Experimental): Patients receive BKM120 PO daily and rituximab IV. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with asymptomatic progression may continue treatment for up to 12 months. Pharmacodynamic samples from peripheral blood (for those with peripheral blood involvement) and bone marrow aspirate (for all patients) are drawn at baseline. Patients will undergo correlative studies to include bone marrow biopsy at study enrollment, and at the time of complete remission.
  Interventions: Drug: PI3K inhibitor BKM120; Biological: rituximab; Other: Pharmacodynamics; Other: Correlative studies

INTERVENTIONS:
Drug: PI3K inhibitor BKM120 — Will be supplied to each patient on the first day of each cycle. It will subsequently be self administered by the patient themselves daily on days 1-28 of every 28 day cycle
  Other Names: BKM120; PI3K_Inhibitor_BKM120
Biological: rituximab — Given IV (intervenously) on days 2, 8, 15, and 22 of cycle 1, and subsequently on day 1 of cycles 3, 5, 7, 9, and 11.
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: Pharmacodynamics — Pharmacodynamic samples from peripheral blood (for those with peripheral blood involvement) and bone marrow aspirate (for all patients) are drawn at baseline.
  Other Names: pharmacological studies; Correlative studies
Other: Correlative studies — Patients will undergo correlative studies to include bone marrow biopsy at study enrollment, and at the time of complete remission. In addition, patients with peripheral blood involvement at enrollment will have peripheral blood drawn for all planned research correlates.
  Other Names: laboratory biomarker analysis

SUMMARY:
This phase I clinical trial studies the side effects and the best dose of phosphatidylinositol-3-kinase (PI3K) inhibitor BKM120 when given together with rituximab in treating patients with relapsed or refractory low-grade B-cell lymphoma. PI3K inhibitor BKM120 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving PI3K inhibitor BKM120 with rituximab may be an effective treatment for B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of combined rituximab and BKM120 (PI3k inhibitor BKM120) in patients with previously treated indolent non-Hodgkin lymphoma (NHL) (including follicular lymphoma (FL), marginal zone lymphoma, and lymphoplasmacytic lymphoma/Waldenstrom's macroglobulinemia), and mantle cell lymphoma (MCL).

SECONDARY OBJECTIVES:

I. To determine specific toxicities associated with combined BKM120 and rituximab.

II. Evaluate for efficacy of BKM120 in combination with rituximab in these diseases.

OUTLINE: This is a dose-escalation study of PI3K inhibitor BKM120.

Patients receive PI3K inhibitor BKM120 orally (PO) daily on days 1-28 and rituximab intravenously (IV) on days 2, 8, 15, and 22 of course 1 and on day 1 of courses 3, 5, 7, 9, and 11. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with asymptomatic progression may continue treatment for up to 12 months.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed indolent B-cell NHL or mantle cell lymphoma; acceptable subtypes of indolent B-cell NHL include follicular lymphoma (grades 1, 2, or 3a), marginal zone lymphoma, or lymphoplasmacytic lymphoma/Waldenstrom's macroglobulinemia; patients with mantle cell lymphoma must have a documented t(11;14) or overexpression of cyclin D1 by immunohistochemical evaluation; patients with active large cell transformation are not eligible; however, patients with a history of large cell transformation are eligible provided that there is no current clinical evidence of active transformed lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least one prior therapy; prior autologous or allogeneic stem cell transplant is allowed; patients may not be on chronic immunosuppressive therapy for graft-versus-host disease (GVHD); patients who have received prior treatment with a pan-selective PI3K inhibitor are not eligible; however, prior therapy with a selective PI3K inhibitor, Bruton's tyrosine kinase inhibitor, or other B-cell receptor targeting agents is allowed
* Serum creatinine =< 2.0 mg/dL
* Total bilirubin =< upper limit of normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.0 x upper limit of normal
* Absolute neutrophil count (ANC) >= 750/mm^3
* Platelets >= 50,000/ mm^3
* Serum lipase =< upper limit of normal
* Serum amylase =< upper limit of normal
* International normalized ratio (INR) =< 2.0
* Fasting glucose < 120mg/dL
* Recovery to =< grade 1 toxicities associated with prior therapy
* Negative serum pregnancy test; if, on cycle 1 day 1, greater than 72 hours has elapsed since the last negative result, a serum pregnancy test must be repeated and be negative on cycle 1 day 1 (C1D1) for the patient to remain eligible
* Patient has the ability and willingness to provide informed consent and has signed the informed consent document

Exclusion Criteria:

* Pregnant or breast-feeding women and women of childbearing age or men who are unwilling to use adequate contraception; females of childbearing age and potential (i.e., not surgically sterilized) must use a second form of contraception, including total abstinence, intra-uterine device, double-barrier contraception, or other non-hormonal form of contraception
* Patients with a history of central nervous system involvement by lymphoma
* The presence of co-existing medical conditions that would limit compliance with study medications, including, but not limited to active infection, active or untreated cardiac or pulmonary disease, or malignancy
* Patients with significant, symptomatic deterioration of lung function confirmed by spirometry, diffusion capacity of carbon monoxide (DLCO), or resting oxygen (O2) saturation
* Patients with impairment of gastrointestinal function that may alter the absorption of BKM120
* Patients currently being actively treated or who have been treated within the past 3 years for an unrelated malignancy (except non-melanoma skin cancer, cervical carcinoma in-situ, and low risk prostate cancer)
* Patients who have undergone major surgery within 2 weeks prior to study enrollment or who have not recovered from a major surgery
* Patients with known human immunodeficiency virus (HIV), hepatitis B or hepatitis C (active or carriers)
* Patients with a fasting blood glucose >= 120 mg/dL (6.7mmol/L); patients with diabetes mellitus are eligible if they require oral agents only and have a fasting blood glucose =< 120 mg/dL; patients with a history of diabetes mellitus who require daily long-acting or mealtime insulin are not eligible; patients who have previously required treatment for hyperglycemia due to steroids or other medications are eligible as long as they have not required insulin or any other oral agent within 2 months prior to study enrollment
* Patients who are on chronic steroids for unrelated conditions (i.e. rheumatologic conditions) are not eligible if their total daily dose of steroids is >= 10mg prednisone
* Patients with a known hypersensitivity to BKM120 or its excipients
* Patients with active moderate or severe major mood or psychiatric disorder as judged by the investigator, primary care physician, counselor, psychiatrist, or as a result of the patient's mood assessment questionnaire that may interfere with the ability to comply with the trial; in addition, given the prior mood-associated toxicities, patients with a history of psychiatric hospitalization within the past 5 years, electroconvulsive therapy (ECT) within the past 5 years, or whose psychiatric condition has been unstable within 2 months prior to study enrollment requiring addition or change of psychotropic medications are not eligible; examples include, but are not limited to:

  * Medically documented history of or active major depressive episode requiring inpatient or intensive outpatient therapy, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or active ideation, or homicidal ideation (immediate risk of doing harm to others); patients under the care of a primary care physician who are treated with one oral agent and who have not required dose adjustments or new medications within 2 months prior to study enrollment and who otherwise meet eligibility requirements may be enrolled
  * >= Common Terminology for Adverse Events (CTCAE) version 4.0 grade 3 anxiety
  * Patients meeting the cutoff score of >= 12 in the Patient Health Questionnaire-9 (PHQ-9) or a cut-off of >= 15 in the Generalized Anxiety Disorder-7 (GAD-7) mood scale, respectively, or who select a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) are not eligible
* Patients with diarrhea >= CTCAE grade 2
* Patients with active cardiac disease including any of the following:

  * Left ventricular ejection fraction < 50% as determined by multi gated acquisition scan (MUGA) scan or echocardiogram
  * Corrected QT interval (QTc) > 480 msec on screening ECG (using the QTcF formula)
  * Active angina pectoris
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular or nodal arrhythmias or any conduction abnormality requiring a pacemaker or automatic implantable cardioverter defibrillator (AICD)
  * Valvular disease with documented compromise in cardiac function
  * Symptomatic pericarditis
  * Myocardial infarction within the past 6 months
  * Congestive heart failure (New York Heart Association [NYHA] functional classification III-IV)
* Patients who are currently receiving treatment with medications with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to study enrollment
* Patients who have taken herbal medications and certain fruits within 7 days prior to study enrollment are not eligible; herbal medications include, but are not limited to, St John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng; exclusionary fruits include the cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A) inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits
* Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to study enrollment; (please note that co-treatment with weak inhibitors of CYP3A is allowed)
* Patients who have received oral or IV chemotherapy, targeted anticancer therapy or radiation therapy =< 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to study enrollment
* Patients who are currently taking therapeutic doses of warfarin sodium or any other Coumadin-derivative anticoagulant; patients who can be safely changed to enoxaparin or other non-warfarin derived anti-coagulant and who otherwise meet eligibility requirements may be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level at which no more than one of 6 patients experiences a DLT summarized using the National Cancer Institute (NCI) CTCAE version 4.0 | 28 days
  Summarized and tabulated by dose level.

SECONDARY OUTCOMES:
Incidence of grade 3 or greater adverse events summarized using the NCI CTCAE version 4.0 | Up to 5 years
  Summarized and tabulated by dose-level.
Overall response rate (ORR) evaluated by computed tomography (CT) or positron emission tomography (PET)/CT | Up to 5 years
Change in correlative markers in blood, bone marrow and tumor tissue | Baseline to up to 5 years
  Explored using graphical analyses as well as summarized quantitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Kami Maddocks, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu